CLINICAL TRIAL: NCT04611737
Title: Developing and Testing of Integrating Self-Determination Theory and Motivational Interviewing Based Diabetic Self-management Program Among Schizophrenic Patients With Diabetes
Brief Title: Self-Determination Theory and Motivational Interviewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMUHIRB-SV(I)-20200019
Record Dates: First submitted 2020-10-25; First posted 2020-11-02 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia; Diabetes
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus | interventions — Interviews as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The researcher interviews with participants for 3 times.
  Interventions: Behavioral: Interviewing
- Control group (No Intervention): The participants receive usual care.

INTERVENTIONS:
Behavioral: Interviewing — Self-Determination Theory within motivational interviewing
  Arms: Experimental group

SUMMARY:
Self-Determination Theory and motivational interviewing would be integrated to enhance the efficacy of diabetic self-management for patients with schizophrenia and Type 2 Diabetes.

DETAILED DESCRIPTION:
Participants would be randomly allocated into either the intervention group or the usual care group from baseline to 3 months follow-up. The intervention is based on integrated self-determination theory and motivational interviewing.

ELIGIBILITY:
Inclusion Criteria:

* patients with schizophrenia and Type 2 Diabetes
* between 20 years old to 80 years old
* can communicate in Chinese langue

Exclusion Criteria:

* can not communicate well
* have neurocognitive disorders

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
HbA1C | on interviewing day1, and 3 months
  Blood sugar level during the 3 months
Body weight | on interviewing day1, and 3 months
  weight (in kilograms)
height | on interviewing day1, and 3 months
  height (in meters), eight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale | on interviewing day1, and 3 months
  The Brief Psychiatric Rating Scale with 18 items is use to measure psychiatric symptoms. Each symptom is rated 1-7 with higher scores indicating severer symptoms.
Treatment Self-Regulation Questionnaire-Diabetes | on interviewing day1, and 3 months
  The treatment Self-Regulation Questionnaire-Diabetes a 19-item scale used to examine the self-regulation behaviors for diabetes of participants. Each item is ranged from 1 to 7 and higher scores showing more motivations in self-regulation diabetes.
Perceived Diabetes Self-Management Scale | on interviewing day1, and 3 months
  The Perceived Diabetes Self-Management Scale is an 8-item scale with 4 of the items (1, 2, 6, & 7) being reverse-scored. Each item is ranged from 1 to 5 and higher scores showing more confidence in self-managing diabetes.
Depression Anxiety Stress Scales | on interviewing day1, and 3 months
  The Depression Anxiety Stress Scales is a self-report scale with 21 items designed to assess depression, stress and anxiety of participants. Scores for each symptom is ranged from 0 to 3 with higher scores indicating severer symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yun Yu, PhD, Principal Investigator — Assistant professor, School of Nursing, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No